CLINICAL TRIAL: NCT05956691
Title: A Phase II, Randomized, Double-blind, Controlled, Single-centre 21-day Study to Investigate the Efficacy of AllerPops to Reduce Nasal Symptoms in Adult Volunteers With Seasonal/Year-long Nasal Allergies
Brief Title: AllerPops Reduce Nasal Symptoms in Adult Volunteers With Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AllerPops Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-SAHSE-01
Record Dates: First submitted 2023-06-16; First posted 2023-07-21 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Allergic Rhinitis
Keywords: allergies; pollen; allergic rhinitis; common allergies; seasonal allergies; yearlong allergies; food allergies; autoimmune; prebiotics; probiotic; natural allergy relief
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity; Rhinitis, Allergic, Seasonal; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigation (Experimental): Dosing Instructions
  1. Brush teeth with water (no toothpaste).
  2. Scrub tongue with warm, wet, washcloth from the back to the front until most of the white/yellow biofilm on the tongue is gone.
  3. Gargle and swish hot (optimal 120°F) water for 10-20 seconds. Spit out and repeat gargling over the next 5 minutes. The tongue should be red and without any biofilm. If it is not, repeat Step 2, and gargle once more.
  4. Self-administer one lozenge. Let the lozenge slowly melt in the mouth. Do not chew or swallow whole. This may take up to 60 minutes. Discard if it is not fully dissolved after 60 minutes.
  5. Wash the washcloth to be ready before next use.
  Interventions: Dietary Supplement: AllerPops
- Control (Active Comparator): Dosing Instructions
  1. Microwave: heat the product in 5 second increments until soft. (Caution: more than 10 seconds of microwaving the product may cause it to burn).
  2. Cut: cut the product into smaller pieces
  3. Swallow: swallow without chewing the pieces with warm water while they are still warm. It can be swallowed over time or at once.
  Interventions: Dietary Supplement: AllerPops

INTERVENTIONS:
Dietary Supplement: AllerPops — Take AllerPops once every other day, as instructed, for a minimum of 3 doses. After each dose, wait at least 30 minutes before eating your next meal. After the 3rd dose, you may continue every other day until you are satisfied with the symptom relief up to and including Day 13.

SUMMARY:
The goal of this clinical trial is to test AllerPops' effectiveness in people who suffer from allergic rhinitis. The main question[s]it aims to answer are:

1. To assess the effectiveness of AllerPops on relieving nasal symptoms compared to the control group in volunteers with seasonal/year-long allergies during the first 7 days of the 21-day intervention period.
2. To evaluate the safety of AllerPops administration in volunteers with seasonal/year-long allergies during a 21-day intervention period.

Up to 30 days between Screening (V1) and Baseline (V2), and a 21-day intervention period, with dosing occurring every other day for a minimum of 3 doses, and thereafter until the participant is satisfied with the relief of the nasal allergy symptoms. The suitable season for the trial will be determined based on the seasonal variation measures.

Researchers will compare slow and fast consuming groups to see if the way of use impact the effectiveness.

DETAILED DESCRIPTION:
Duration: Up to 30 days between Screening (V1) and Baseline (V2), and a 21-day intervention period, with dosing occurring every other day for a minimum of 3 doses, and thereafter until the participant is satisfied with the relief of the nasal allergy symptoms. The suitable season for the trial will be determined based on the seasonal variation measures.

Primary Objectives: To assess the effectiveness of AllerPops on relieving nasal symptoms compared to the control group in volunteers with seasonal/year-long allergies during the first 7 days of the 21-day intervention period.

Secondary Objective:

1. To evaluate the safety of AllerPops administration in volunteers with seasonal/year-long allergies during a 21-day intervention period.
2. To assess the duration of effectiveness of AllerPops in relieving nasal symptoms compared to the control group in volunteers with seasonal/year-long allergies during a 21-day intervention period (exploratory).
3. To evaluate the effect of the AllerPops administration on the oral microbial presentation/microbiota using Amplicon Metagenomics Sequencing test through saliva samples during a 21-day intervention period (exploratory).
4. To evaluate the effect of the AllerPops administration on the IgE (total) blood level during a 21-day intervention period (exploratory).

Study Population: Seventy-two participants with seasonal/year-long nasal allergies.

Duration: Up to 30 days between Screening (V1) and Baseline (V2), and a 21-day intervention period, with dosing occurring every other day for a minimum of 3 doses, and thereafter until the participant is satisfied with the relief of the nasal allergy symptoms. The suitable season for the trial will be determined based on the seasonal variation measures.

Primary Objectives: To assess the effectiveness of AllerPops on relieving nasal symptoms compared to the control group in volunteers with seasonal/year-long allergies during the first 7 days of the 21-day intervention period.

Secondary Objective:

1. To evaluate the safety of AllerPops administration in volunteers with seasonal/year-long allergies during a 21-day intervention period.
2. To assess the duration of effectiveness of AllerPops in relieving nasal symptoms compared to the control group in volunteers with seasonal/year-long allergies during a 21-day intervention period (exploratory).
3. To evaluate the effect of the AllerPops administration on the oral microbial presentation/microbiota using Amplicon Metagenomics Sequencing test through saliva samples during a 21-day intervention period (exploratory).
4. To evaluate the effect of the AllerPops administration on the IgE (total) blood level during a 21-day intervention period (exploratory).

Study Population: Seventy-two participants with seasonal/year-long nasal allergies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participants will be clinically diagnosed with persistent or intermittent allergic rhinitis, according to the Allergic Rhinitis and Its Impact on Asthma (ARIA) classification. (The guidelines of Allergic Rhinitis and its Impact on Asthma (ARIA) group, classified it to intermittent (less than 4 days per week and for less than 4 weeks) and persistent (more than 4 days per week or lasting more than 4 weeks regardless of the number of days per week).

  2. Male or female seasonal/year-long nasal allergy sufferers (as assessed by a questionnaire at screening) between the ages of 18 and 70.

  3. Females who are not of childbearing potential (post-menopausal defined as those with amenorrhea for at least 2 years). Females of childbearing potential should be either sexually inactive (abstinent) for 60 days prior to the first dose of the study, throughout the study and for 30 days after completion of the study, or be using one of the following acceptable methods of birth control: i. Surgically sterile (bilateral tubal-ligation, hysterectomy, bilateral oophorectomy) for at least 90 days prior to the first dose of the study.

ii. IUD in place for at least 60 days prior to the first dose of the study, throughout the study and for 30 days after completion of the study.

iii. Barrier methods (condom, diaphragm) with spermicide for at least 60 days prior to the first dose of the study, throughout the study and for 30 days after study completion.

iv. Hormonal contraceptives for at least 90 days prior to the first dose of the study, throughout the study, and for 30 days after study completion.

* Changes to the method of birth control while participating in the study will be judged by the PI for acceptability.

  4. Written informed consent obtained and signed by participant. 5. BMI between 18.5 and 29.9 kg/m2, with a stable weight over the last 3 months. (A stable weight is defined as <5% of total body weight change in the last 3 months).

  6. Agrees not to use any over the counter, prescription, health supplement or dietary supplement from at least 14 days prior to screening until the end of the study.

  7. Agrees to maintain current dietary habits, level of physical activity, occupational and living environment for the trial duration.

  8. Does not regularly consume more than 2 standard* alcoholic beverages a day as assessed through verbal confirmation at screening, and agrees not to consume >2 standard* alcoholic beverages per day for the trial duration.

  9. Non-smoker within 12 months prior to dosing as assessed by verbal confirmation.

  10. Stable medical conditions that do not require medication use routinely and do not affect or involve the immune systems as determined by medical history, physical examination, clinical chemistry performed at screening, and as assessed by the Principal Investigator.

  11. Agrees not to use nasal steroid spray from at least 14 days prior to screening until the end of the study.

  12. Agrees not to use neti-pot and oil-pulling for at least 7 days prior to screening until the end of the study.

  13. . 14. Have access to a microwave.

Exclusion Criteria:

1. Participants who are pregnant/lactating or planning to become pregnant during the course of the clinical trial.
2. Participants who have any sings of active or recurrent upper airway infection (bacterial/viral).
3. Participants who have a known sensitivity or allergy to any of the study products, or ingredients.
4. Participation in another research study within 30 days prior to enrollment in this clinical trial.
5. Participants who are not able to tolerate venipuncture and/or have poor venous access.
6. Participants dependent on decongestants (nasal or oral) or receiving allergen-specific immunotherapy.
7. Participants who have been diagnosed with other clinical forms of rhinitis such as infectious rhinitis, rhinitis of pregnancy, food and alcohol-induced rhinitis, atrophic rhinitis, vasomotor rhinitis, rhinosinusitis and age-related rhinitis.
8. Participants who have receive previous acupuncture treatment or alternative medicine for AR in the last three months or planned in the next two years.
9. Participants who have received allergy desensitization therapy (current, during the past two years, or planned in the next two years).
10. Participants who have had any major surgery within 1 year of enrollment into the clinical trial or have any anticipated major surgeries intended to occur during the clinical trial.
11. Participants who have received a blood transfusion within 8 weeks of enrollment in the clinical trial.
12. Participants who have donated blood or plasma to a blood bank or clinical study within 8 weeks of enrollment and during the study except venipuncture as part of clinical trial.
13. Participant has known severe medical conditions, such as cardiovascular, liver or renal dysfunction, diabetes mellitus, cancers, cerebrovascular diseases, blood system diseases which in the opinion of the Principal Investigator, may preclude safe study participation, or interfere with study objectives.
14. Participants who are immunocompromised or have been diagnosed HIV/AIDS, Hepatitis B, or untreated Hepatitis C.
15. Participant has a history of alcohol or drug addiction treatment within the last 2 years prior to inclusion in the study, or any current addiction on alcohol or drugs.
16. Participants with Grade II or III septum deviation and/or presence of nasal polyps or other conditions that lead to nasal obstruction.
17. Participant has any other medical, social or other condition that, in the opinion of the Principal Investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
18. Participants with allergic asthma and/or moderate to severe atopic dermatitis.
19. History of anaphylactic reactions.
20. Participants with any risk of developing dental cavity or on-going oral health issue, as assessed during their regular dentist visit in past 6 months.
21. Participants who brush more than twice a day and/or mouthwash more than once a day and/or floss more than once a day.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Allergy symptom changes measured by severity grade (0-3) in TNSS(Total Nasal Symptoms Score) Questionnaire. | 21-day
  To assess the effectiveness of AllerPops on changing nasal symptoms in volunteers with seasonal/year-long allergies during the first 7 days of the 21-day intervention period.
  Total Nasal Symptoms Score (TNSS) Questionnaire in grades of 0-3: a method developed to assess allergic rhinitis symptoms, based on the administration of a questionnaire. According to this method, allergic rhinitis symptoms are scored from 0 to 3 (4 grades of severity). This assessment will be conducted at the D1, D7, D14 and D21.
Nasal air flow changes measured by liter per minute in PNIF (Peak Nasal Inspiratory Flow) measurement. | 21-day
  To assess the effectiveness of AllerPops on altering nasal air flow in volunteers with seasonal/year-long allergies during the first 7 days of the 21-day intervention period.
  Peak Nasal Inspiratory Flow (PNIF) measured in liter per minute: Measures nasal flow for assessing nasal airway patency. This assessment will be conducted at the D1, D7, D14 and D21.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by monitoring of vital signs, complete blood count, and a comprehensive safety panel. | 21 days
  To evaluate the safety of AllerPops administration in volunteers with seasonal/year-long allergies during a 21-day intervention period.
  a. Safety will be assessed by collecting vital signs (temperature, blood pressure, heart rate), the emergence of adverse events, and clinical chemistry (complete blood count, CBC [Includes: White Blood Cell Count (WBC), Red Blood Cell Count (RBC), Hemoglobin (HB), Hematocrit (HCT), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), and mean corpuscular hemoglobin concentration (MCHC), Platelet Count] and a comprehensive safety panel: Aspartate aminotransferase (AST), Sodium, Potassium, Chloride, Serum creatinine, Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Bilirubin Total and Gamma Glutamyl Transpeptidase (GGT)), and PI assessment.
  This assessment will be conducted at the baseline D1, D7, D14 and D21.
Changes in participants' oral microbiomes using 16S amplicon metagenomic sequencing. | 21 days
  The exploratory study of the effect of AllerPops in oral microbial presentation/microbiota through Amplicon Metagenomics Sequencing test which is a rRNA gene (V3-V4 region) sequencing method in saliva. The evaluation will be measured at D1, D7 and D21.

CONTACTS AND LOCATIONS:
Overall Officials: Raj Gurinder, MD, Principal Investigator — Independent
Locations (1):
- Dicentra, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shunsheng Han C. Prebiotic supplements correct oral probiotic deficiency for lasting allergy relief. Am J Transl Res. 2024 Jan 15;16(1):136-146. doi: 10.62347/JWOU4205. eCollection 2024. PMID 38322553

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05956691/Prot_SAP_000.pdf